CLINICAL TRIAL: NCT05350527
Title: Impact of a Personalized and Secure Video Information Support and Web Platform on Preoperative Anxiety in the Context of Breast Cancer Surgery
Brief Title: Impact of Video Information Support on Preoperative Anxiety in Breast Cancer Surgery
Acronym: SENEDOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: EDOP Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RECHMPL21_0680
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Preoperative Anxiety; Preoperative information; Video support; Web platform; Breast cancer surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the clinical research associate (CRA) will know the patient's arm. The rest of the clinical team will be blinded. The self-questionnaires will be completed by the patients and then retrieved by the CRA who will enter the data into the eCRF, with no possible access to this data by the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Web platform and video information support (Experimental): After usual preoperative information delivered by surgeon, patients allocated to Arm will be able to access to video information support and web platform.
  Interventions: Other: Consultation of a Web Platform
- Arm B: Standard Preoperative information (No Intervention): Patients randomized in Arm B will only receive usual preoperative information delivered by the surgeon.

INTERVENTIONS:
Other: Consultation of a Web Platform — Patients willing to participate in this research and randomized in the experimental arm will benefit, in addition to standard preoperative medical information, an access to the EDOP internet platform via personalized and secure access codes. They will be able to watch an explanatory video about breast surgery and find all the essential, practical and useful information about their intervention and the postoperative effects for the duration of their follow-up.
  Arms: Arm A: Web platform and video information support

SUMMARY:
The medical information delivered to the patient before any surgery constitutes an essential and compulsory step during the initial management of the operated patient.

There are different reasons for the quantity and quality of medical information retained by the patient. An internet platform with personalized and secure access has been developed. This platform contains, among other things, an explanatory video of breast surgery and allows the patient to have access to information on surgical management at any time.

The investigators believe that unlimited access for the duration of the study to this platform could reduce the preoperative anxiety level of patients.

DETAILED DESCRIPTION:
The medical information provided during the pre-operative phase is an essential and mandatory step in the duty to inform during the initial management of the patient undergoing surgery. The different reasons acting on the quantity and quality of the medical information integrated by the patient can be linked to several factors: among others, the information supports, the age, the listening and comprehension capacities, the level of anxiety or the level of education of the patient, thus creating health inequalities. The use of visual communication seems to be more suitable for patients with a low level of education, illiteracy or non-native speakers. Studies have shown that, in addition to oral preoperative information, the introduction of a visual medium with the use of a video has demonstrated a significant reduction in preoperative anxiety and the use of the Internet.

The prevalence of anxiety is high in cancer patients, particularly during the preoperative phase. The EDOP company has developed a personalized and secure Internet platform containing, among other things, an explanatory video on breast surgery. In the current literature, there are no studies on the contribution of the use of video and web platform in the context of preoperative medical information.

In this study, the investigators hypothesize that the unlimited access to the EDOP platform and the possibility to review as many times as necessary the information concerning their surgical intervention could allow, whatever the situation of the patients, to reduce the level of preoperative anxiety, which is always deleterious. Indeed, studies have shown the negative effects of preoperative anxiety on the quantity of anaesthetic used during the operation or on the consumption of analgesics postoperatively. A reduction in preoperative anxiety would therefore be likely to lead in the short term to a reduction in drug treatments and probably to a better state of health.

The main objective is to evaluate the impact of additional personalized preoperative medical information, accessible via a secure internet platform, on anxiety on the morning of surgery, in the context of breast cancer surgery, after conventional oral and written information.

The secondary objectives are to compare between the 2 groups:

* the change in anxiety between the preoperative visit and the morning of the procedure,
* patient satisfaction and understanding of the preoperative medical information received after the preoperative visit, on the morning of the operation, at discharge (between D0 and D3) and at the postoperative visit (6 weeks),
* consultation of other websites and contact with the medical team, on the morning of the operation and at the post-operative visit (6 weeks),
* the quantity of anaesthetic products used during the operation
* the consumption of analgesics during the 15 days after the operation
* consumption of anxiolytics during the 15 postoperative days

For the experimental group:

* To evaluate the use of the EDOP platform,
* To evaluate patient satisfaction with this platform.

This is a Multicenter, prospective, randomized, single-blind study. Only the clinical study technician (CST) will know the patient's group. Nursing staff will be blinded. Self-questionnaires will be filled out by the patients and then retrieved by the CT who will enter the data into the eCRF, with no access to these data by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast cancer.
* Indication of breast lumpectomy, oncoplasty or mastectomy.
* Person over 18 years old

Exclusion Criteria:

* Person with a history of breast cancer surgery.
* Person with severely impaired physical and/or psychological health, which, in the opinion of the investigator, may affect the participant's compliance to the study.
* Individuals who have difficulty understanding the French language orally.
* Person who does not have Internet access at home or at work.
* Person placed under court protection.
* Person who is not a member or beneficiary of a national health insurance system.
* Person who has not given oral informed consent after a reflection period.
* Person participating in another research study with an exclusion

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with perioperative anxiety symptoms | The morning of surgery (Day 0)
  Anxiety is assessed with the Amsterdam Preoperative Anxiety and Information Scale (APAIS) using 3 distinct areas: Anesthesia Anxiety (items 1 and 2), Surgery Anxiety (items 4 and 5), and Need for Information (items 3 and 6).Each question is measured on a 5-point scale ranging from 1 "not at all" to 5 "extremely". To obtain the overall anxiety score, the scores of the 4 anxiety items (1, 2, 4 and 5) are added together. Subjects are considered anxious when they have a score strictly higher than 10 for these 4 items.

SECONDARY OUTCOMES:
Evolution of anxiety related to the surgery | The pre-operative consultation and the morning of the surgery (Day 0)
  The evolution of anxiety related to the surgery is evaluated by the variation on score of the Amsterdam Preoperative Anxiety and Information Scale (APAIS) between the preoperative consultation and the morning of the intervention.
  The APAIS using 3 distinct areas: Anesthesia Anxiety (items 1 and 2), Surgery Anxiety (items 4 and 5), and Need for Information (items 3 and 6).Each question is measured on a 5-point scale ranging from 1 "not at all" to 5 "extremely". To obtain the overall anxiety score, the scores of the 4 anxiety items (1, 2, 4 and 5) are added together. Subjects are considered anxious when they have a score strictly higher than 10 for these 4 items.
Evaluation of satisfaction and understanding of preoperative medical information | The pre-operative consultation, the morning of the surgery (Day 0), at discharge (between Day 0 and 3) and at the postoperative visit (at 6 weeks)
  This outcome is evaluated by the Medical Information Comprehension and Satisfaction Assessment Questionnaire was designed to assess 3 items: quality of medical information, comprehension of different topics, and overall satisfaction with medical information.
  To calculate the score:
  * items are rated from 1 (Not at all) to 5 (Totally) for questions 1 and 3
  * items are rated from 5 (Not at all) to 1 (Totally) for question 2
  * Visual Analogue Scale: 1 point for a score of 0 to 20, 2 points for a score of 21 to 40, 3 points for a score of 41 to 60, 4 points for a score of 61 to 80, 5 points for a score of 81 to 100 (question 4).
Rate of patients who used the Internet and/or contacted the gynecology department | The morning of the surgery (Day 0) and at the postoperative visit (at 6 weeks)
  The Questionnaire evaluating Internet use and contact with the gynecology department was designed to assess the use of the Internet and contact with the clinical team to obtain additional information about the procedure. It also assesses the reasons for using or not using the Internet, as well as the reliability of the information consulted on the Internet.
  The patient must specify whether she consults the Internet in a general way for her health (item 1) and she must indicate whether or not she has used the internet since the last visit to obtain additional information about her procedure (item 2), she must give:
  * If yes, the reasons for using the Internet (items 3, 4 and 5)
  * If no, the reasons for not using the Internet (items 6) The patient must mention whether she contacted the gynecology department by phone and/or email (item 7) and whether she consulted urgently for her breast surgery (item 8), in order to obtain additional information about the procedure.
Intravenous anesthetic consumption | Day of the surgery (Day 0)
  The consumption of intravenous anesthetic is mesured by the hypnotics in milligrams and morphine in micrograms. This data will be collected from the patient's computerized medical record.
Use of analgesics | 15 postoperative days
  Use of analgesics is classified in 3 categories: levels 1, 2 and 3. A calendar will be given to patients so that they can record their use of analgesics during the 15 days postoperatively. This calendar will be retrieved at the 6-week postoperative visit
Number of days of use of anxiolytics | 15 postoperative days
  A calendar will be given to patients so that they can record their use of anxiolytics during the 15 days postoperatively. This calendar will be retrieved at the 6-week postoperative visit
Number of connections to the EDOP platform for experimental group | The morning of the surgery (Day 0) and at the post-operative visit (at 6 weeks)
  The number of connections to the EDOP platform is assessed for patients in the experimental group (Arm A), using question 1 of the questionnaire evaluating the number of connections and patient satisfaction with the EDOP platform.
Satisfaction of the experimental group | The morning of the surgery (Day 0) and at the post-operative visit (at 6 weeks)
  The satisfaction of the patients in the experimental group is assessed using the questionnaire evaluating the number of connections and the satisfaction of the patients concerning the EDOP platform (Questions 3, 7 and 8)

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, MD, Study Director — Montpellier University Hospital
Locations (4):
- France (4):
  - CH Béziers, Béziers
  - Clinique de Clémentville, Montpellier
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No